CLINICAL TRIAL: NCT04028024
Title: Study on the Protective Effect of Inhibiting Systemic Inflammatory Response in Patients Undergoing Cardiac Surgery.
Brief Title: Protective Effect in Cardiac Surgery Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B2019-156
Record Dates: First submitted 2019-07-14; First posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Cardiac Surgery
MeSH Terms: interventions — urinastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- inhibiting systemic inflammatory response (Other): Ulinastatin 5000U/kg in 20ml NS i.v. before occlusion of aorta
  Interventions: Drug: Ulinastatin

INTERVENTIONS:
Drug: Ulinastatin — Ulinastatin 5000U/Kg in 20 ml NS i.v. before occlusion of aorta

SUMMARY:
The purpose of the study was to verify the protective effect of inhibiting systemic inflammatory response in patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* subject needs to have valve surgery
* subject needs to have coronary artery bypass grafting surgery
* subject needs to have artificial blood vessel replacement surgery
* ASA(American Society of Anesthesiologists) score II~III
* NYHA(New York Heart Association) II~III

Exclusion Criteria:

* LVEF(left ventricular ejection fraction) <40% measured by echocardiogram
* history of myocardial infarction within 1 month
* history of serious pulmonary infection or endocarditis within 3 months
* history of important surgery within 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
postoperative delirium | 7 days postoperatively or discharge, whichever came first
  the incidence of postoperative delirium
postoperative renal insufficiency | 7 days postoperatively or discharge, whichever came first
  the incidence of renal insufficiency

CONTACTS AND LOCATIONS:
Overall Officials: Hui-lin Wang, Phd, Principal Investigator — Fudan University